CLINICAL TRIAL: NCT00591084
Title: Efficacy and Safety of Ginsenoside-Rd for Acute Ischemic Stroke: A Randomized, Double-blind, Placebo-controlled, Phase Ⅱ, Multicenter Trial
Brief Title: Ginsenoside-Rd for Acute Ischemic Stroke
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: the neurology department of Xijing Hospital, Xijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: xijing-001
Record Dates: First submitted 2007-12-27; First posted 2008-01-11 (Estimated); Last update posted 2010-09-01 (Estimated); Status verified 2007-12

CONDITIONS: Ischemic Stroke
Keywords: randomized trial; ischemic stroke; Ginsenoside-Rd
MeSH Terms: conditions — Ischemic Stroke | interventions — ginsenoside Rd

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ginsenoside-Rd 10mg (Experimental): both a ginsenoside-Rd injection (10mg/1ml/each) and a specific dilution (10%, 1ml trimethylene glycol) were respectively diluted by a specific dilution (10%, 9 ml trimethylene glycol) and then mixed.
  Interventions: Drug: ginsenoside-Rd 10 mg
- placebo (Placebo Comparator): 2 specific dilutions (10%, 1ml trimethylene glycol) were respectively diluted by 2 specific dilutions (10%, 9 ml trimethylene glycol) and then mixed.
  Interventions: Drug: placebo
- ginsenoside-Rd 20mg (Experimental): 2 ginsenoside-Rd injections (10mg/1ml/each) were respectively diluted by 2 specific dilutions (10%, 9 ml trimethylene glycol) and then mixed
  Interventions: Drug: ginsenoside-Rd 20mg

INTERVENTIONS:
Drug: ginsenoside-Rd 10 mg — infusion ginsenoside-Rd 10 mg (group A)once a day and continued for 14 days
  Arms: ginsenoside-Rd 10mg
Drug: placebo — infusion placebo (group B)once a day and continued for 14 days
  Arms: placebo
Drug: ginsenoside-Rd 20mg — infusion of ginsenoside-Rd 20mg (group C) once a day and continued for 14 days
  Arms: ginsenoside-Rd 20mg

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of ginsenoside-Rd for acute ischemic stroke.

DETAILED DESCRIPTION:
A major contributor to brain injury after stroke is disordered inward flow of Ca2+ and its toxic accumulation in the nervous system following cerebral ischemia. Ginsenoside-Rd, a purified component from total saponins of Panax notoginseng, has a molecular formula of C48H82O18•3H2O with a molecular weight of 1001.2. Ginsenoside-Rd has been shown to inhibit receptor-operated Ca2+ influx through receptor-and-store-operated Ca2+ channels (ROCC) , attenuate oxidative stress in stroke, reduce the size of the cerebral infarction and preserve brain functioning in animal models of acute ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* between 18 to 75 years
* the first episode
* from onset to admission within 72 hours
* NIHSS scores:5~22

Exclusion Criteria:

* had other intracranial pathologies (e.g., tumor, infection)
* had a neurologic or psychiatric disease
* had a coexisting condition that limited their life expectancy
* had significant drug or alcohol misuse
* had high-grade carotid artery stenosis for which surgery was planned
* were pregnant or nursing
* participated in a clinical trial with an investigational drug or device within the past 3 months
* were unlikely to be available for follow-up

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2005-09; Primary Completion 2006-06 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
NIHSS scores | 15±1 days

SECONDARY OUTCOMES:
NIHSS scores | 8 days
the Barthel index | 8 days
the Barthel index | 15 days
the modified Rankin scale | 15 days
the modified Rankin scale | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Gang Zhao, MD, Study Director — the Department of Neurology , Xijing Hospital;; Xuedong Liu, MD, Study Chair — the Department of Neurology, Xijing Hospital;
Locations (1):
- the Department of Neurology , Xijing Hospital, Xi'an, Shaanxi, China

REFERENCES:
- [Derived] Liu X, Xia J, Wang L, Song Y, Yang J, Yan Y, Ren H, Zhao G. Efficacy and safety of ginsenoside-Rd for acute ischaemic stroke: a randomized, double-blind, placebo-controlled, phase II multicenter trial. Eur J Neurol. 2009 May;16(5):569-75. doi: 10.1111/j.1468-1331.2009.02534.x. Epub 2009 Feb 19. PMID 19236467